CLINICAL TRIAL: NCT04573699
Title: BackBeat Medical Cardiac Neuromodulation Therapy in Patients With Heart Failure: An Acute Feasibility Study
Brief Title: Cardiac Neuromodulation for Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BackBeat Medical Inc (Industry)
Collaborators: CD Leycom (Unknown)
Responsible Party: Sponsor
Other Study IDs: BBM HF-CS-01
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CNT-HF — A modified CNT, will be delivered as a pacing sequence able to acutely influence sympathetic tone.

SUMMARY:
This investigation will evaluate the ability of the Moderato® System to safely and effectively deliver CNT, to reduce sympathetic activity in heart failure patients

DETAILED DESCRIPTION:
This will be a single center, non-randomized observational study. The Moderato® System is approved for marketing in Europe (has a CE mark) for the treatment of high blood pressure in patients requiring standard cardiac pacing. The therapy delivered by the Moderato® System is referred to as CNT (Cardiac Neuromodulation Therapy). Heart failure patients is a population for which the Moderato® device is currently not indicated.

Subjects requiring an implantable cardiac defibrillator (ICD) implantation or replacement and meeting study inclusion and exclusion criteria will be eligible to participate in the study. The study procedure will take place during the ICD implantation (or replacement).

The whole procedure will be performed according to standard of care for ICD implantations (or replacements) including periprocedural prophylactic antibiotics prophylactic. To reduce the time of wound exposure, the setup of system for invasive measurements will be done before the ICD implant (or replacement) procedure begins.

The groin area will be prepared and draped. After applying local anesthesia, a 7Fr sheath will be inserted into the femoral artery. A small dose of heparin (~5000 units) will be administered intravenously to prevent formation of blood clots. Under fluoroscopic guidance, a standard conductance catheter (CD Leycom CA-71103-PL, CE marked) will be advanced into the left ventricle.

The arterial line will be used to measure arterial pressure. This completes the measuring system setup.

Then, ICD right atrial lead and right ventricular lead will be implanted in standard positions according to standard institutional practices.

The leads will be connected to a BackBeat Moderato® System IPG, externally to the patient using a single use, sterile Pacing System Analyzer (PSA) cable provided by the hospital. The Moderato® IPG, approved for chronic CNT delivery in hypertensive patients, will function in this trial as a temporary external CNT signal generator for acute application of the therapy.

A range of CNT signal parameters will be used to assess the effect on sympathetic activity. Ventricular pressure and volume readings from the conductance catheter and arterial pressure readings will be recorded and analyzed to assess the effect of CNT signals on cardiac function, sympathetic activity and blood pressure. The effects of CNT signal over a range of parameter settings will be studied over a period of time no longer than one hour.

In this study, none of the Moderato® system components will be in contact with the patient. The Moderato® IPG will be used solely as an external CNT signal generator and deliver signals to the patient through the PSA cable and the ICD leads.

When CNT signal activation is complete, data recording will be stopped, the conductance catheter will be removed, the cable connecting the IPG to the leads disconnected, and ICD implantation will proceed normally.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject has a primary indication and is scheduled for ICD implantation or replacement
3. Subject has heart failure NYHA Class II or III

Exclusion Criteria:

1. Subject is to receive a single chamber defibrillator
2. Subject has an ejection fraction of 25% or less
3. Subject's systolic blood pressure is less than 120 mm Hg on the day of implant
4. Subject has decompensated heart failure
5. Subject has significant (>2+) mitral regurgitation, aortic regurgitation or aortic stenosis.
6. Subject has permanent atrial fibrillation
7. Subject has atrial fibrillation on the day of the study.
8. Subject has hypertrophic cardiomyopathy, restrictive cardiomyopathy or interventricular septal thickness ≥15 mm
9. Subject has a history of prior neurological events (stroke or TIA) within the past year or a neurological event (stroke or TIA) at any prior time that has resulted in residual neurologic deficit.
10. Subject has a history of autonomic dysfunction
11. Women who are pregnant or breast-feeding
12. Subject cannot or is unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are Heart Failure subjects willing to participate in a short acute clinical study during the implantation or replacement of a single chamber ICD.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Arterial Elastance | Immediate, derived form ongoing Pressure Volume changes in the Left ventricle
  Arterial elastance is reduced when sympathetic activity is reduced, an indication of a relaxed peripheral resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Kalarus, Prof. MD Ph.D, Principal Investigator — Silesian Center for Heart Diseases
Locations (1):
- Silesian Center for Heart Diseases, Zabrze, Poland

REFERENCES:
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the diagnosis and treatment of acute and chronic heart failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur J Heart Fail. 2008 Oct;10(10):933-89. doi: 10.1016/j.ejheart.2008.08.005. Epub 2008 Sep 16. No abstract available. PMID 18826876
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):188-97. doi: 10.1161/CIR.0b013e3182456d46. No abstract available. PMID 22215894
- [Background] van Bilsen M, Patel HC, Bauersachs J, Bohm M, Borggrefe M, Brutsaert D, Coats AJS, de Boer RA, de Keulenaer GW, Filippatos GS, Floras J, Grassi G, Jankowska EA, Kornet L, Lunde IG, Maack C, Mahfoud F, Pollesello P, Ponikowski P, Ruschitzka F, Sabbah HN, Schultz HD, Seferovic P, Slart RHJA, Taggart P, Tocchetti CG, Van Laake LW, Zannad F, Heymans S, Lyon AR. The autonomic nervous system as a therapeutic target in heart failure: a scientific position statement from the Translational Research Committee of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2017 Nov;19(11):1361-1378. doi: 10.1002/ejhf.921. Epub 2017 Sep 26. PMID 28949064